CLINICAL TRIAL: NCT04660643
Title: Efficacy and Safety of Tirzepatide Once Weekly Versus Placebo for Maintenance of Weight Loss in Participants Without Type 2 Diabetes Who Have Obesity or Are Overweight With Weight-Related Comorbidities: A Randomized, Double-Blind, Placebo-Controlled Trial (SURMOUNT-4)
Brief Title: A Study of Tirzepatide (LY3298176) in Participants With Obesity or Overweight for the Maintenance of Weight Loss
Acronym: SURMOUNT-4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17247; I8F-MC-GPHN (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-12-01; First posted 2020-12-09 (Actual); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Obesity; Overweight
Keywords: Metabolism and Nutrition Disorder; Prediabetes
MeSH Terms: conditions — Obesity; Overweight; Nutrition Disorders; Prediabetic State | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tirzepatide (lead-in) (Experimental): Participants received weekly doses of tirzepatide subcutaneously (SC) for 36 weeks, starting at 2.5 milligrams (mg) and increasing by 2.5 mg every 4 weeks, as tolerated, up to the maximum tolerated dose (MTD) of either 10 mg or 15 mg.
  Interventions: Drug: Tirzepatide
- Tirzepatide MTD (Experimental): Participants continued tirzepatide MTD (either 10 mg or 15 mg) for an additional 52 weeks.
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Participants received weekly doses of placebo SC for 52 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Tirzepatide (lead-in); Tirzepatide MTD
Other: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
This was a study of tirzepatide in participants with obesity or overweight. The main purpose was to learn more about how tirzepatide maintained body weight loss. The study had two phases: a lead-in phase in which all participants took tirzepatide and a treatment phase in which participants either continued tirzepatide or switched to placebo. The study lasted about 2 years (25 visits).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥30 kilograms per square meter (kg/m²), or ≥27 kg/m² and previous diagnosis with at least one of the following comorbidities: hypertension, dyslipidemia, obstructive sleep apnea, cardiovascular disease
* History of at least one unsuccessful dietary effort to lose body weight

Exclusion Criteria:

* Diabetes mellitus
* Change in body weight greater than 5 kg within 3 months prior to starting study
* Obesity induced by other endocrinologic disorders or monogenetic or syndromic forms of obesity
* History of pancreatitis
* Family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2)
* History of significant active or unstable major depressive disorder (MDD) or other severe psychiatric disorder within the last 2 years
* Any lifetime history of a suicide attempt

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 783 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (70):
- United States (48):
  - Cahaba Research, Pelham, Alabama
  - Scripps Memorial Hospital La Jolla, La Jolla, California
  - National Research Institute - Wilshire, Los Angeles, California
  - National Research Institute, Panorama City, California
  - Artemis Institute for Clinical Research, San Diego, California
  - University Clinical Investigators, Inc., Tustin, California
  - New West Physicians Clinical Research, Golden, Colorado
  - Optumcare Colorado Springs - Monument, Monument, Colorado
  - Care Partners Clinical Research, Jacksonville, Florida
  - South Florida Clinical Research Institute, Margate, Florida
  - Renstar Medical Research, Ocala, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - SKY Clinical Research Network Group-Blake, Union City, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Healthcare Research Network - Chicago, Flossmoor, Illinois
  - Clinical Investigation Specialists, Gurnee, Illinois
  - Midwest Institute For Clinical Research, Indianapolis, Indiana
  - American Health Network of Indiana, LLC - New Albany, New Albany, Indiana
  - Cotton O'Neil Clinic, Topeka, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Centennial Medical Group, Elkridge, Maryland
  - MedStar Health Research Institute (MedStar Physician Based Research Network), Hyattsville, Maryland
  - ActivMed Practices and Research, Methuen, Massachusetts
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Glacier View Research Institute - Endocrinology, Kalispell, Montana
  - Weill Cornell Medical College, New York, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - Wake Forest University Baptist Medical Center (WFUBMC), Winston-Salem, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - Aventiv Research Inc, Columbus, Ohio
  - Intend Research, LLC, Norman, Oklahoma
  - Summit Research Network, Portland, Oregon
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - The University of Texas Health Science Center at Houston, Bellaire, Texas
  - Dallas Diabetes Research Center, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - North Hills Family Medicine/North Hills Medical Research, North Richland Hills, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Northwest Houston Heart Center, Tomball, Texas
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - Capital Clinical Research Center, Olympia, Washington
  - Rainier Clinical Research Center, Renton, Washington
- Argentina (7):
  - CEDIC, CABA, Buenos Aires
  - Centro Médico Viamonte, CABA, Buenos Aires
  - Stat Research S.A., Ciudad Autónoma de Buenos Aire, Buenos Aires
  - Mautalen Salud e Investigación, Buenos Aires, Ciudad Autónoma de Buenos Aire
  - Centro Medico Dr Laura Maffei Investigacion Clinica Aplicada, Ciudad Autonoma de Buenos Aire, Ciudad Autónoma de Buenos Aire
  - Instituto Médico Catamarca IMEC, Rosario, Santa Fe Province
  - Asociación de Beneficencia Hospital Sirio Libanés, Buenos Aires
- Brazil (8):
  - CEDOES, Vitória, Espírito Santo
  - Cline Research Center, Curitiba, Paraná
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Sao Lucas, Campinas, São Paulo
  - ISPEM - Instituto São José dos Campos em Pesquisas Médicas, São José dos Campos, São Paulo
  - BR Trials - Ensaios Clinicos e Consultoria, São Paulo, São Paulo
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - CPQuali Pesquisa Clínica, São Paulo
- Puerto Rico (3):
  - Centro de Endocrinologia Alcantara Gonzalez, Bayamón
  - Private Practice Dr. Martha Gomez Cuellar, San Juan
  - Wellness clinical Research Vega Baja, Vega Baja
- Taiwan (4):
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - National Cheng-Kung Uni. Hosp., Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Almandoz JP, Pickett-Blakely O, Tewksbury C, Stefanski A, Gonsahn-Bollie S, Dimitriadis GK, Murro AL, Cao D, Meng Q, Neff LM. Nutritional status with tirzepatide in obesity: A post hoc analysis of the SURMOUNT-1-4 randomized clinical trials. Obes Pillars. 2026 Jan 23;17:100248. doi: 10.1016/j.obpill.2026.100248. eCollection 2026 Mar. PMID 41640675
- [Derived] Horn DB, Linetzky B, Davies MJ, Laffin LJ, Wang H, Murphy MA, Zimner-Rapuch S, Lau E, Arad AD, Lee CJ. Cardiometabolic Parameter Change by Weight Regain on Tirzepatide Withdrawal in Adults With Obesity: A Post Hoc Analysis of the SURMOUNT-4 Trial. JAMA Intern Med. 2025 Nov 24:e256112. doi: 10.1001/jamainternmed.2025.6112. Online ahead of print. PMID 41284285
- [Derived] Li X, Cao D, Sapin H, Wang F, Hunter Gibble T, Raibulet NK, Denning M, Kaplan LM. People With Lowest Physical Functioning Scores Showed Greatest Improvement After Tirzepatide Treatment. Obesity (Silver Spring). 2026 Jan;34(1):114-126. doi: 10.1002/oby.70067. Epub 2025 Nov 4. PMID 41187013
- [Derived] Gibble TH, Cao D, Murphy M, Jouravskaya I, Liao B, Bays HE. Tirzepatide Associated With Improved Health-Related Quality of Life in Adults With Obesity or Overweight in SURMOUNT-4. Obesity (Silver Spring). 2025 Nov;33(11):2076-2092. doi: 10.1002/oby.70011. Epub 2025 Sep 3. PMID 40903801
- [Derived] Gourgari E, Srivastava G, Kelly AS, Mojdami D, Cao D, Murphy MA, Karanikas CA, Lee CJ. Early-Onset Obesity and Tirzepatide Treatment: A Post Hoc Analysis of the SURMOUNT Clinical Trials. Obesity (Silver Spring). 2025 Sep;33(9):1668-1679. doi: 10.1002/oby.24348. Epub 2025 Jul 27. PMID 40717199
- [Derived] Horn DB, Kahan S, Batterham RL, Cao D, Lee CJ, Murphy M, Gonsahn-Bollie S, Chigutsa F, Stefanski A, Dunn JP. Time to weight plateau with tirzepatide treatment in the SURMOUNT-1 and SURMOUNT-4 clinical trials. Clin Obes. 2025 Jun;15(3):e12734. doi: 10.1111/cob.12734. Epub 2025 Jan 12. PMID 39800653
- [Derived] Aronne LJ, Sattar N, Horn DB, Bays HE, Wharton S, Lin WY, Ahmad NN, Zhang S, Liao R, Bunck MC, Jouravskaya I, Murphy MA; SURMOUNT-4 Investigators. Continued Treatment With Tirzepatide for Maintenance of Weight Reduction in Adults With Obesity: The SURMOUNT-4 Randomized Clinical Trial. JAMA. 2024 Jan 2;331(1):38-48. doi: 10.1001/jama.2023.24945. PMID 38078870
- See also: A Study of Tirzepatide (LY3298176) in Participants With Obesity or Overweight for the Maintenance of Weight Loss (SURMOUNT-4) — https://trials.lillytrialguide.com/en-US/trial/aK2GGZSCqbdJMNUlhfAVV

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: * Open-label lead-in period: Baseline (week 0) to week 36: Participants received weekly doses of tirzepatide SC escalated every 4 weeks until they attained a maximum tolerated dose (MTD).
  * Double-blind study period (randomized period including the safety follow-up): Randomization (week 36) to week 92: At week 36, those who completed the lead-in treatment were randomized 1:1 to tirzepatide MTD and placebo, treated up to week 88, and followed up for safety after 4 weeks off treatment, at week 92.
Period: Open-label Lead-in Period (Week 0 - 36)
Arm/Group | Tirzepatide (lead-in) | Placebo | Tirzepatide MTD
Started | 783 | 0 | 0
Received at Least 1 Dose of Study Drug | 782 | 0 | 0
Completed 36-weeks of Treatment (i.e., Reaching and Tolerating the MTD at Week 36) (Eligible for randomization.) | 670 | 0 | 0
Completed (All enrolled participants with a non-missing body weight measurement at week 36, regardless of treatment discontinuation were considered as lead-in period completers.) | 671 | 0 | 0
Not Completed | 112 | 0 | 0
Not completed — Adverse Event | 50 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 14 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol deviation | 10 | 0 | 0
Not completed — Withdrawal by Subject | 32 | 0 | 0
Not completed — Covid-19 | 1 | 0 | 0
Not completed — Other - as reported by the investigator | 2 | 0 | 0
Period: Double-blind Study Period (Week 36 - 92)
Arm/Group | Tirzepatide (lead-in) | Placebo | Tirzepatide MTD
Started | 0 (Lead-in period arm.) | 335 (Randomized arm.) | 335 (Randomized arm.)
Received at Least 1 Dose of Study Drug | 0 | 335 | 335
Completed | 0 | 290 | 310
Not Completed | 0 | 45 | 25
Not completed — Death | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 10 | 8
Not completed — Pregnancy | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 22 | 13
Not completed — Protocol deviation | 0 | 1 | 2
Not completed — Other - as reported by the investigator | 0 | 8 | 0
Not completed — Perceived excessive weight loss | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tirzepatide MTD | Total
Number analyzed (Participants) | 335 | 335 | 670
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.15 (12.38) | 48.27 (12.79) | 47.71 (12.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 237 | 236 | 473
  Male | 98 | 99 | 197
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 155 | 141 | 296
  Not Hispanic or Latino | 180 | 193 | 373
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 22 | 26 | 48
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 36 | 39 | 75
  White | 273 | 264 | 537
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 56 | 55 | 111
  Brazil | 46 | 43 | 89
  Taiwan | 17 | 21 | 38
  United States | 216 | 216 | 432
Body weight [Mean (Standard Deviation); unit: kilogram (kg)] | 107.79 (23.66) | 106.82 (20.94) | 107.3 (22.33)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Randomization in Body Weight at Week 88
Description: Least square (LS) mean was analysed by mixed model repeated measures (MMRM) model with randomization + analysis country + sex + interactive web response system (IWRS) MTD at Week 36 + treatment + time + treatment*time (Type III sum of squares) as variables.
Time Frame: Randomization (Week 36), Week 88
Population: All randomized participants who received at least one dose of the study drug, had randomization and at least one post-randomization values for this outcome, excluding data after discontinuation of the study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 329 | 332
percent change | 14.8 (0.53) | -6.7 (0.52)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -21.4, 95% CI 2-sided [-22.9 to -20.0]

2. Secondary Outcome: Percent Change From Randomization in Body Weight at Week 64
Description: LS mean was analysed by MMRM model with randomization + analysis country + sex + IWRS MTD at Week 36 + treatment + time + treatment*time (Type III sum of squares) as variables.
Time Frame: Randomization (Week 36), Week 64
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 329 | 332
percent change | 9.9 (0.38) | -6.0 (0.37)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -15.9, 95% CI 2-sided [-17.0 to -14.9]

3. Secondary Outcome: Change From Randomization in Body Weight
Description: as for outcome 2
Time Frame: Randomization (Week 36), Week 88
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 329 | 332
kilogram (kg) | 11.9 (0.43) | -5.7 (0.42)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -17.6, 95% CI 2-sided [-18.8 to -16.4]

4. Secondary Outcome: Change From Randomization in Waist Circumference
Description: LS mean was analysed by MMRM model with randomization + analysis country + sex + IWRS MTD at Week 36 + weight loss at week 36 (< 10%, >= 10%) + treatment + time + treatment*time (Type III sum of squares) as variables.
Time Frame: Randomization (Week 36), Week 88
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: centimetre (cm)
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 329 | 332
centimetre (cm) | 8.3 (0.44) | -4.6 (0.43)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -12.9, 95% CI 2-sided [-14.1 to -11.7]

5. Secondary Outcome: Change From Randomization in Body Mass Index (BMI)
Description: as for outcome 2
Time Frame: Randomization (Week 36), Week 88
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilogram per square metre (kg/m^2)
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 329 | 332
kilogram per square metre (kg/m^2) | 4.3 (0.16) | -2.1 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -6.4, 95% CI 2-sided [-6.8 to -6.0]

6. Secondary Outcome: Change From Randomization in Fasting Glucose
Description: as for outcome 4
Time Frame: Randomization (Week 36), Week 88
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 310 | 325
milligrams per deciliter (mg/dL) | 7.74 (0.548) | -0.90 (0.528)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -8.64, 95% CI 2-sided [-10.14 to -7.15]

7. Secondary Outcome: Change From Randomization in Hemoglobin A1c (HbA1c)
Description: as for outcome 4
Time Frame: Randomization (Week 36), Week 88
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 311 | 325
percentage of HbA1c | 0.25 (0.017) | -0.08 (0.017)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -0.33, 95% CI 2-sided [-0.38 to -0.28]

8. Secondary Outcome: Percent Change From Randomization in Fasting Insulin
Description: LS mean was analysed by MMRM model with log(actual measurement/randomization) = log (randomization) + analysis country + sex + IWRS MTD at Week 36 + weight loss at week 36 (< 10%, >= 10%) + treatment + time + treatment*time (Type III sum of squares) as variables.
Time Frame: Randomization (Week 36), Week 88
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 311 | 324
percent change | 23.3 (4.37) | -15.4 (2.88)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -31.4, 95% CI 2-sided [-37.7 to -24.4], Standard Error of Mean 3.37

9. Secondary Outcome: Percent Change From Randomization in Lipid Parameters (Total Cholesterol, Low Density Lipoprotein (LDL) Cholesterol, High Density Lipoprotein (HDL) Cholesterol, Very Low Density Lipoprotein (VLDL) Cholesterol, Triglycerides, Free Fatty Acids (FFA))
Description: as for outcome 8
Time Frame: Randomization (Week 36), Week 88
Population: All randomized participants who received at least one dose of the study drug, had randomization and at least one post-randomization values for the respective lipid parameters, excluding data after discontinuation of the study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 273 | 298
percent change
  Total Cholesterol | 8.30 (0.943) | 2.29 (0.852)
  LDL Cholesterol: number analyzed (Participants) | 270 | 297
  LDL Cholesterol | 3.43 (1.368) | -3.36 (1.218)
  HDL Cholesterol: number analyzed (Participants) | 272 | 298
  HDL Cholesterol | 14.6 (1.06) | 18.3 (1.05)
  VLDL Cholesterol: number analyzed (Participants) | 268 | 297
  VLDL Cholesterol | 14.7 (2.32) | -7.8 (1.77)
  Triglycerides: number analyzed (Participants) | 270 | 297
  Triglycerides | 15.6 (2.39) | -8.2 (1.81)
  FFA: number analyzed (Participants) | 264 | 291
  FFA | -2.9 (2.98) | -13.4 (2.54)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Total Cholesterol; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -5.54, 95% CI 2-sided [-7.76 to -3.28], Standard Error of Mean 1.139
Statistical Analysis 2: Comparison: Placebo vs Tirzepatide MTD; LDL Cholesterol; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -6.57, 95% CI 2-sided [-9.87 to -3.15], Standard Error of Mean 1.709
Statistical Analysis 3: Comparison: Placebo vs Tirzepatide MTD; HDL Cholesterol; Test type: Superiority; p = 0.014, Mixed Models Analysis; LS Mean difference = 3.2, 95% CI 2-sided [0.6 to 5.8], Standard Error of Mean 1.33
Statistical Analysis 4: Comparison: Placebo vs Tirzepatide MTD; VLDL Cholesterol; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -19.7, 95% CI 2-sided [-24.0 to -15.1], Standard Error of Mean 2.25
Statistical Analysis 5: Comparison: Placebo vs Tirzepatide MTD; Triglycerides; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -20.6, 95% CI 2-sided [-24.9 to -16], Standard Error of Mean 2.27
Statistical Analysis 6: Comparison: Placebo vs Tirzepatide MTD; FFA; Test type: Superiority; p = 0.008, Mixed Models Analysis; LS Mean difference = -10.8, 95% CI 2-sided [-17.9 to -3.0], Standard Error of Mean 3.79

10. Secondary Outcome: Change From Randomization in Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP)
Description: LS mean change was analysed by MMRM model with randomization + analysis country + sex + IWRS MTD at Week 36 + Weight Loss at Week 36 (< 10%, >= 10%) + treatment + time + treatment*time (Type III sum of squares) as variables.
Time Frame: Randomization (Week 36), Week 88
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimetre of mercury (mmHg)
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 329 | 332
millimetre of mercury (mmHg)
  SBP | 8.4 (0.64) | 2.1 (0.61)
  DBP | 3.2 (0.44) | -0.4 (0.42)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; SBP; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -6.4, 95% CI 2-sided [-8.1 to -4.6]
Statistical Analysis 2: Comparison: Placebo vs Tirzepatide MTD; DBP; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -3.6, 95% CI 2-sided [-4.8 to -2.4]

11. Secondary Outcome: Change From Randomization in Short Form 36 Version 2 Health Survey (SF 36v2) Acute Form - Physical Functioning Domain Score
Description: The SF-36v2 acute form assesses health-related quality of life (HRQoL) on 8 domains: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. The Physical-Functioning domain assesses limitations due to health "now" and consists of 10-items, each rated on a 3-point Likert scale. Scoring of the domain is norm-based and presented in the form of T-scores, with a mean of 50 and standard deviation of 10; higher scores indicate better levels of function. Range cannot be specified in norm-based scores.
  LS mean was analysed by analysis of covariance (ANCOVA) model with randomization + analysis Country + sex + weight loss at Week 36 (< 10%, >= 10%) + IWRS MTD at Week 36 + treatment (type III sum of squares) as variables.
Time Frame: Randomization (Week 36), Week 88
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 270 | 295
T-score | -1.8 (0.32) | 0.8 (0.31)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Test type: Superiority; p < .001, ANCOVA; LS Mean difference = 2.6, 95% CI 2-sided [1.7 to 3.5]

12. Secondary Outcome: Change From Randomization in Impact of Weight on Quality of Life Lite Clinical Trials Version (IWQOL-Lite-CT) - Physical Function Composite Score
Description: The IWQOL Lite-CT consists of 20 items, assessing 2 primary domains of obesity related HRQoL: Physical (7 items) and Psychosocial (13 items). A 5-item subset of the Physical domain - the Physical Function composite - is also supported. Items in the Physical Function composite describe physical impacts related to general and specific physical activities. All items in the physical domain are rated on either a 5-point frequency ("never" to "always") scale or a 5-point truth ("not at all true" to "completely true") scale. Total score of IWQOL-Lite-CT composite ranges from 0 to 100, with higher scores reflecting better health-related quality of life.
  LS mean was analysed by ANCOVA model with randomization + analysis Country + sex + weight loss at Week 36 (< 10%, >= 10%) + IWRS MTD at Week 36 + treatment (type III sum of squares) as variables.
Time Frame: Randomization (Week 36), Week 88
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 272 | 293
score on a scale | -5.0 (0.95) | 4.4 (0.91)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference = 9.4, 95% CI 2-sided [6.8 to 12.0]

13. Secondary Outcome: Percentage of Participants Who Maintain at Least 80% of the Body Weight Lost During the Open-Label Lead-In Period
Description: Percentage of Participants Who Maintain at least 80% of the Body Weight Lost During the Open-Label Lead-In Period was analysed by Logistic regression model with missing value imputed by MMRM at week 88. Missing values were imputed by predictions using observed data in the efficacy analysis set from the same treatment group through an MMRM analysis model for post-baseline measures with Baseline + Analysis Country + Sex + IWRS MTD at Week 36 + randomization + Treatment + Time + Treatment*Time as variables.
Time Frame: Week 88
Population: All randomized participants who received at least one dose of the study drug, had weight loss in the open label lead-in period and at least one post-randomization value for this outcome, excluding data after discontinuation of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 326 | 332
percentage of participants | 13.50 | 93.37
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 95.91, 95% CI 2-sided [54.72 to 168.09]

14. Secondary Outcome: Percentage of Participants Who Achieve ≥5%, ≥10%, ≥15%, ≥20% Body Weight Reduction From Baseline
Description: Percentage of Participants Who Achieve ≥5%, ≥10%, ≥15%, ≥20% Body Weight Reduction from baseline was analysed by Logistic regression model with missing value imputed by MMRM at week 88. Missing values were imputed by predictions using observed data in the efficacy analysis set from the same treatment group through an MMRM analysis model for post-baseline measures with Baseline + Analysis Country + Sex + IWRS MTD at Week 36 + randomization + Treatment + Time + Treatment*Time as variables.
Time Frame: Baseline (Week 0) to Week 88
Population: All randomized participants who received at least one dose of the study drug, had baseline and at least one post-randomization values for this outcome, excluding data after discontinuation of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 329 | 332
percentage of participants
  ≥5% body weight reduction from baseline | 69.00 | 98.49
  ≥10% body weight reduction from baseline | 44.38 | 93.98
  ≥15% body weight reduction from baseline | 24.01 | 87.05
  ≥20% body weight reduction from baseline | 11.55 | 72.59
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; ≥5% body weight reduction from baseline; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 47.27, 95% CI 2-sided [18.32 to 121.99]
Statistical Analysis 2: Comparison: Placebo vs Tirzepatide MTD; ≥10% body weight reduction from baseline; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 71.51, 95% CI 2-sided [34.46 to 148.39]
Statistical Analysis 3: Comparison: Placebo vs Tirzepatide MTD; ≥15% body weight reduction from baseline; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 79.99, 95% CI 2-sided [42.06 to 152.14]
Statistical Analysis 4: Comparison: Placebo vs Tirzepatide MTD; ≥20% body weight reduction from baseline; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 140.84, 95% CI 2-sided [66.06 to 300.29]

15. Secondary Outcome: Time to First Occurrence of Participants Returning to >95% Baseline Weight for Those Who Lost ≥5% During the Open-Label Lead-In Period
Description: Time to first occurrence of participants returning to >95% baseline weight for those who lost ≥5% during the open-label lead-in period.
Time Frame: Randomization (Week 36) to Week 88
Population: All randomized participants who received at least one dose of the study drug, lost >=5% of their weight in the open label period, excluding data after discontinuation of study drug.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 327 | 332
weeks | NA [NA to NA] — There were not enough events to estimate the median and confidence interval. | NA [NA to NA] — There were not enough events to estimate the median and confidence interval.
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Test type: Superiority; p < .001, Log Rank; Hazard Ratio (HR) = 0.013, 95% CI 2-sided [0.004 to 0.046] — Unstratified hazard ratio from Cox proportional hazard model with Baseline Weight (kg), Analysis Country, Sex, IWRS MTD at Week 36, Weight at randomization (kg) as covariates

16. Secondary Outcome: Change From Baseline in BMI
Description: LS mean was analysed by MMRM model with baseline + analysis country + sex + IWRS MTD at Week 36 + BMI at randomization (kg/m^2) + treatment + time + treatment*time (Type III sum of squares) as variables.
Time Frame: Baseline (Week 0), Week 88
Population: All randomized participants who received at least one dose of the study drug, had baseline and at least one post-baseline values for this outcome, excluding data after discontinuation of the study drug.
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 329 | 332
kg/m^2 | -3.6 (0.16) | -10.0 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -6.4, 95% CI 2-sided [-6.8 to -6.0]

17. Secondary Outcome: Change From Baseline in Body Weight
Description: LS mean was analysed by MMRM model with baseline + analysis country + sex + IWRS MTD at Week 36 + body weight at randomization (kg) + treatment + time + treatment*time (Type III sum of squares) as variables.
Time Frame: Baseline (Week 0), Week 88
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 329 | 332
kg | -10.0 (0.43) | -27.6 (0.42)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -17.6, 95% CI 2-sided [-18.8 to -16.4]

18. Secondary Outcome: Percent Change From Baseline in Body Weight
Description: as for outcome 17
Time Frame: Baseline (Week 0), Week 88
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 329 | 332
percent change | -9.5 (0.40) | -26.0 (0.39)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -16.4, 95% CI 2-sided [-17.5 to -15.4]

19. Secondary Outcome: Change From Baseline in Waist Circumference
Description: LS mean was analysed by MMRM model with baseline + analysis country + sex + IWRS MTD at Week 36 + weight loss at week 36 (< 10%, >= 10%) + treatment + time + treatment*time (Type III sum of squares) as variables.
Time Frame: Baseline (Week 0), Week 88
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 329 | 332
cm | -9.1 (0.53) | -22.8 (0.52)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -13.6, 95% CI 2-sided [-15.1 to -12.2]

20. Secondary Outcome: Change From Baseline in Fasting Glucose
Description: as for outcome 19
Time Frame: Baseline (Week 0), Week 88
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 310 | 325
mg/dL | -1.72 (0.543) | -10.63 (0.522)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -8.92, 95% CI 2-sided [-10.40 to -7.43]

21. Secondary Outcome: Change From Baseline in HbA1c
Description: as for outcome 19
Time Frame: Baseline (Week 0), Week 88
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 311 | 325
percentage of HbA1c | -0.22 (0.018) | -0.57 (0.017)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -0.34, 95% CI 2-sided [-0.39 to -0.29]

22. Secondary Outcome: Percent Change From Baseline in Fasting Insulin
Description: LS mean was analysed by MMRM model with log(actual measurement/baseline) = log (baseline) + analysis country + sex + IWRS MTD at Week 36 + weight loss at week 36 (< 10%, >= 10%) + treatment + time + treatment*time (Type III sum of squares) as variables.
Time Frame: Baseline (Week 0), Week 88
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 300 | 314
percent change | -29.8 (2.52) | -54.1 (1.57)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -34.6, 95% CI 2-sided [-40.6 to -27.9], Standard Error of Mean 3.25

23. Secondary Outcome: Percent Change From Baseline in Lipid Parameters (Total Cholesterol, LDL Cholesterol, HDL Cholesterol, VLDL Cholesterol, Triglycerides, FFAs)
Description: as for outcome 22
Time Frame: Baseline (Week 0), Week 88
Population: All randomized participants who received at least one dose of the study drug, had baseline and at least one post-baseline values for the respective lipid parameters, excluding data after discontinuation of the study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 273 | 298
percent change
  Total Cholesterol | 2.16 (0.919) | -5.01 (0.817)
  LDL Cholesterol: number analyzed (Participants) | 270 | 297
  LDL Cholesterol | 2.62 (1.371) | -5.21 (1.207)
  HDL Cholesterol: number analyzed (Participants) | 272 | 298
  HDL Cholesterol | 9.44 (1.093) | 12.29 (1.071)
  VLDL Cholesterol: number analyzed (Participants) | 266 | 297
  VLDL Cholesterol | -15.6 (1.82) | -32.6 (1.37)
  Triglycerides: number analyzed (Participants) | 270 | 297
  Triglycerides | -15.3 (1.84) | -33.3 (1.38)
  FFA: number analyzed (Participants) | 264 | 291
  FFA | -9.69 (2.811) | -20.38 (2.360)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Total Cholesterol; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -7.02, 95% CI 2-sided [-9.27 to -4.72], Standard Error of Mean 1.158
Statistical Analysis 2: Comparison: Placebo vs Tirzepatide MTD; LDL Cholesterol; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -7.62, 95% CI 2-sided [-10.91 to -4.21], Standard Error of Mean 1.707
Statistical Analysis 3: Comparison: Placebo vs Tirzepatide MTD; HDL Cholesterol; Test type: Superiority; p = 0.064, Mixed Models Analysis; LS Mean difference = 2.60, 95% CI 2-sided [-0.14 to 5.43], Standard Error of Mean 1.418
Statistical Analysis 4: Comparison: Placebo vs Tirzepatide MTD; VLDL Cholesterol; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -20.1, 95% CI 2-sided [-24.7 to -15.3], Standard Error of Mean 2.38
Statistical Analysis 5: Comparison: Placebo vs Tirzepatide MTD; Triglycerides; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -21.2, 95% CI 2-sided [-25.8 to -16.4], Standard Error of Mean 2.38
Statistical Analysis 6: Comparison: Placebo vs Tirzepatide MTD; FFA; Test type: Superiority; p = 0.004, Mixed Models Analysis; LS Mean difference = -11.83, 95% CI 2-sided [-18.98 to -4.06], Standard Error of Mean 3.793

24. Secondary Outcome: Change From Baseline in SBP, DBP
Description: as for outcome 19
Time Frame: Baseline (Week 0), Week 88
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 329 | 332
mmHg
  SBP | -2.4 (0.66) | -9.3 (0.63)
  DBP | -1.7 (0.46) | -5.5 (0.44)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; SBP; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -6.9, 95% CI 2-sided [-8.7 to -5.1]
Statistical Analysis 2: Comparison: Placebo vs Tirzepatide MTD; DBP; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean difference = -3.8, 95% CI 2-sided [-5.1 to -2.6]

25. Secondary Outcome: Change From Baseline in SF 36v2 Acute Form - Physical Functioning Domain Score
Description: as for outcome 11
Time Frame: Baseline (Week 0), Week 88
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 271 | 296
T-score | 3.7 (0.36) | 6.3 (0.34)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Test type: Superiority; p < .001, ANCOVA; LS Mean difference = 2.7, 95% CI 2-sided [1.7 to 3.7]

26. Secondary Outcome: Change From Baseline in IWQOL-Lite-CT - Physical Function Composite Score
Description: The IWQOL Lite-CT consists of 20 items, assessing 2 primary domains of obesity related HRQoL: Physical (7 items) and Psychosocial (13 items). A 5-item subset of the Physical domain - the Physical Function composite - is also supported. Items in the Physical Function composite describe physical impacts related to general and specific physical activities. All items in the physical domain are rated on either a 5-point frequency ("never" to "always") scale or a 5-point truth ("not at all true" to "completely true") scale. Total score of IWQOL-Lite-CT composite ranges from 0 to 100, with higher scores reflecting better health-related quality of life.
  LS mean was analysed by ANCOVA model with baseline + analysis Country + sex + weight loss at Week 36 (< 10%, >= 10%) + IWRS MTD at Week 36 + treatment (type III sum of squares) as variables.
Time Frame: Baseline (Week 0), Week 88
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Tirzepatide MTD
Number analyzed (Participants) | 273 | 294
score on a scale | 16.7 (1.01) | 26.0 (0.97)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide MTD; Test type: Superiority; p < .001, ANCOVA; LS Mean difference = 9.3, 95% CI 2-sided [6.5 to 12.0]

ADVERSE EVENTS:
Time Frame: Week 0 to 36 for the open-label lead-in period arm, Week 36 to 92 for the double-blind study period arms.
Description: All participants who received at least one dose of the study drug. Based on the planned safety analysis, adverse events were collected per the treatment regimen, irrespective of dose.
Groups:
- Tirzepatide (lead-in): Participants received weekly doses of tirzepatide SC for 36 weeks, starting at 2.5 mg and increasing by 2.5 mg every 4 weeks, as tolerated, up to the MTD of either 10 mg or 15 mg.
Arm/Group | Tirzepatide (lead-in) | Placebo | Tirzepatide MTD
All-Cause Mortality (participants affected / at risk) | 1/782 | 1/335 | 1/335
Serious Adverse Events (participants affected / at risk) | 16/782 | 10/335 | 10/335
Other Adverse Events (participants affected / at risk) | 559/782 | 100/335 | 124/335
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tirzepatide (lead-in) (N=782) | Placebo (N=335) | Tirzepatide MTD (N=335)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Cholecystitis acute (Hepatobiliary disorders) | 4 (4) | 3 (3) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Aortic aneurysm repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tirzepatide (lead-in) (N=782) | Placebo (N=335) | Tirzepatide MTD (N=335)
Abdominal pain (Gastrointestinal disorders) | 48 (71) | 6 (9) | 11 (12)
Constipation (Gastrointestinal disorders) | 162 (202) | 8 (9) | 12 (17)
Diarrhoea (Gastrointestinal disorders) | 165 (329) | 16 (21) | 36 (112)
Dyspepsia (Gastrointestinal disorders) | 63 (78) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 69 (90) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 278 (600) | 9 (11) | 27 (75)
Vomiting (Gastrointestinal disorders) | 128 (275) | 4 (7) | 18 (36)
Fatigue (General disorders) | 53 (61) | 2 (2) | 9 (12)
Injection site reaction (General disorders) | 64 (424) | 2 (4) | 7 (107)
Covid-19 (Infections and infestations) | 82 (83) | 50 (51) | 47 (47)
Upper respiratory tract infection (Infections and infestations) | 26 (28) | 18 (18) | 8 (9)
Decreased appetite (Metabolism and nutrition disorders) | 74 (145) | 4 (7) | 7 (14)
Headache (Nervous system disorders) | 56 (72) | 10 (10) | 5 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 40 (40) | 5 (5) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT04660643/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT04660643/SAP_001.pdf